CLINICAL TRIAL: NCT01793428
Title: Predictive Abilities for Transfusion Needs of Capillary Lactate Measure in Emergency for Injured Normotensive Patients
Brief Title: Capillary Lactate and Transfusion Needs
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 2012-19
Record Dates: First submitted 2013-02-12; First posted 2013-02-15 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-04

CONDITIONS: Trauma
Keywords: adults admitted in vital emergency unit
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Injured patient admitted in vital emergency unit
  Interventions: Other: Capillary lactate level

INTERVENTIONS:
Other: Capillary lactate level — Use of capillary sample to determine lactate level upon arrival at vital emergency unit and at 2 hours

SUMMARY:
13% of injured normotensive patients arriving in emergency unit need mass blood-transfusion of six or more units of packed Red Blood Cells. It is currently difficult to predict the need for such a mass blood-transfusion. Indeed hemoglobin point of care testing (hemocue) and blood pressure can be normal during the first hours despite intensive bleeding.

It's well known that blood or arterial lactate measures correlate with trauma severity but these measures are not available in a pre-hospital setting. The investigators want to test whether capillary lactate measures also correlate with trauma severity and can therefore predicts earlier transfusion needs.

ELIGIBILITY:
Inclusion Criteria:

* Adult admitted in vital emergency unit
* Severe trauma
* normotensive (Systolic Blood Pressure >90mmHg)
* patient subjected to capillary haemoglobin and glucose measurements
* patient beneficiary of social security

Exclusion Criteria:

* pregnant woman
* liver deficiency
* pre-hospital transfusion
* hypothermia below 35°C
* protected persons according to the law
* Nor epinephrine > 0.1gamma/kg/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults admitted in vital emergency unit due to severe trauma based on a local severity score.
  Patients are normotensive
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2011-08; Primary Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Transfusion of 6 or more units of packed Red Blood Cells (RBC) | 48 hours

SECONDARY OUTCOMES:
arterial lactate measures | upon arrival at the vital emergency unit
injury scores (ISS,SOFA) | 24h
transfusion of 4 units of packed RBC | 48 hours
blood lactate measure | upon arrival at vital emergency unit
Intensity of medical care | upon arrival at vital emergency unit
  Body scan Central venous catheterisation arterial catheterisation
Bleeding Predictive Score | upon arrival at vital emergency unit
  3 questions are asked to the doctor in emergency room. Could patient be admitted directly at the CT scan ? Do you think that the patient need transfusion ? If Yes : and how many units ? Do you think that the patient will be hospitalized in an intensive care unit after the emergency room?
Mortality | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Marc Vinclair, MD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Grenoble University Hospital, La Tronche, Isere, France

REFERENCES:
- [Derived] Bouzat P, Schilte C, Vinclair M, Manhes P, Brun J, Bosson JL, Payen JF. Capillary lactate concentration on admission of normotensive trauma patients: a prospective study. Scand J Trauma Resusc Emerg Med. 2016 Jun 7;24:82. doi: 10.1186/s13049-016-0272-x. PMID 27267942